CLINICAL TRIAL: NCT04968782
Title: Appendicitis Choice of Treatment Study
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, David Flum, Director Surgical Outcomes Research Center, University of Washington
Other Study IDs: STUDY00013390
Record Dates: First submitted 2021-07-08; First posted 2021-07-20 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Acute Appendicitis
Keywords: Decision Making; Decisional Conflict
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with acute appendicitis
  Interventions: Other: Patients with acute appendicitis

INTERVENTIONS:
Other: Patients with acute appendicitis — No intervention, single survey

SUMMARY:
A longitudinal observational/survey study evaluating patient centered decision making in the choice of treatment for acute appendicitis. Survey evaluates patients experience with decision making and the types of decision support they receive.

ELIGIBILITY:
Inclusion Criteria:

* English Speaking
* Diagnosed with acute appendicitis
* Considered by the treating clinical team to be eligible for treatment with surgery or with non operative treatment (antibiotics)
* Access to an internet connected device capable of taking the survey

Exclusion Criteria:

* Patients who do not make their own medical decisions
* Patients who are not felt to be candidates for a decision between operative and nonoperative treatment by the treating clinical team
* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the emergency department with acute appendicitis who are considered to be candidates for operative or nonoperative management by the treating clinical team. Patients can ultimately have undergone either treatment.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2022-02-16 (Actual)

PRIMARY OUTCOMES:
Decisional conflict | Time of survey (2 days-2 weeks after treatment for acute appendicitis)
  Validated evaluation of decision making

SECONDARY OUTCOMES:
Preparation for decision making | Time of survey (2 days-2 weeks after treatment for acute appendicitis)
  Validated measure for patient subject preparedness to make a treatment decision

CONTACTS AND LOCATIONS:
Overall Officials: David R Flum, MD, MPH, Study Director — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Decisional Conflict Scale — https://decisionaid.ohri.ca/eval_dcs.html